CLINICAL TRIAL: NCT00265330
Title: 26-Week Open-Label Extension Study Evaluating The Safety And Tolerability Of Flexible Doses Of Oral Ziprasidone In Children And Adolescents With Bipolar I Disorder (Manic Or Mixed)
Brief Title: Safety and Tolerability of Ziprasidone in Children and Adolescents With Bipolar I Disorder (Manic or Mixed)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A1281133
Record Dates: First submitted 2005-12-12; First posted 2005-12-14 (Estimated); Results first posted 2009-04-03 (Estimated); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Bipolar Disorder
Keywords: Children And Adolescents With Bipolar I Disorder (Manic Or Mixed)
MeSH Terms: conditions — Bipolar Disorder | interventions — ziprasidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open (Experimental)
  Interventions: Drug: Ziprasidone oral capsules

INTERVENTIONS:
Drug: Ziprasidone oral capsules — Study medications will include oral ziprasidone capsules of 20 mg, 40 mg, 60 mg, and 80 mg strength. Subjects will be dosed daily for 26 weeks using a flexible dose design with a minimal dose range of 20mg bid to a maximum dose range of 80 mg bid .

SUMMARY:
The purpose of this study is to assess the safety and tolerability of ziprasidone during long-term open-label administration in children and adolescents (ages 10-17) with bipolar I disorder (manic or mixed)

ELIGIBILITY:
Inclusion Criteria:

* Participation in double-blind treatment study A1281132, meeting specific criteria of duration and safety

Exclusion Criteria:

* Imminent risk of suicide or homicide, as judged by the site investigator;serious adverse event related to study medication in study A1281132; significant prolongation of QT interval in study A1281132.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 169 (Actual)
Dates: Start 2006-03; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (36):
- United States (36):
  - Pfizer Investigational Site, Scottsdale, Arizona
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Altamonte Springs, Florida
  - Pfizer Investigational Site, Fort Lauderdale, Florida
  - Pfizer Investigational Site, North Miami, Florida
  - Pfizer Investigational Site, Orange City, Florida
  - Pfizer Investigational Site, Tavares, Florida
  - Pfizer Investigational Site, Decatur, Georgia
  - Pfizer Investigational Site, Honolulu, Hawaii
  - Pfizer Investigational Site, Terre Haute, Indiana
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Owensboro, Kentucky
  - Pfizer Investigational Site, Shreveport, Louisiana
  - Pfizer Investigational Site, Clinton Township, Michigan
  - Pfizer Investigational Site, Meridian, Mississippi
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Lincoln, Nebraska
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Tulsa, Oklahoma
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Arlington, Texas
  - Pfizer Investigational Site, DeSoto, Texas
  - Pfizer Investigational Site, Lake Jackson, Texas
  - Pfizer Investigational Site, Plano, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Kirkland, Washington
  - Pfizer Investigational Site, Spokane, Washington
  - Pfizer Investigational Site, Milwaukee, Wisconsin
  - Pfizer Investigational Site, West Allis, Wisconsin

REFERENCES:
- [Derived] Findling RL, Cavus I, Pappadopulos E, Vanderburg DG, Schwartz JH, Gundapaneni BK, DelBello MP. Efficacy, long-term safety, and tolerability of ziprasidone in children and adolescents with bipolar disorder. J Child Adolesc Psychopharmacol. 2013 Oct;23(8):545-57. doi: 10.1089/cap.2012.0029. Epub 2013 Oct 10. PMID 24111980
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1281133&StudyName=Safety%20and%20tolerability%20of%20ziprasidone%20in%20children%20and%20adolescents%20with%20bipolar%20I%20disorder%20%28manic%20or%20mixed%29

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The number of subjects entering this trial was determined by the number of subjects electing to continue treatment after completing or withdrawing from the preceding double-blind study (A1281132: NCT00257166).
Pre-assignment Details: A total of 169 subjects from the parent study were assigned to the extension study and 162 continued on and received study treatment in the extension study.
Groups:
- Ziprasidone: Dosing was flexible, with dosing adjustments made at the discretion of the investigator to maintain optimal efficacy and tolerability. For subjects having a body weight of 45 kilograms (kg) or greater, the target dosage range was 40-80 milligrams (mg) twice per day (BID) (80-160 mg/day). For subjects having a body weight under 45 kg, the maximum permitted dose was 80 mg/day (40 mg BID).
Period: Overall Study
Arm/Group | Ziprasidone
Started | 162
Completed | 67
Not Completed | 95
Not completed — Adverse Event | 41
Not completed — Lost to Follow-up | 8
Not completed — Withdrawal by Subject | 34
Not completed — Patient Wanted to Start Psychotherapy | 1
Not completed — Lack of Efficacy | 4
Not completed — Family Scheduling Conflicts | 1
Not completed — Began Taking Formulary Geodon | 1
Not completed — Discharged from Unit for Long Term Care | 1
Not completed — Site Closed by Sponsor | 1
Not completed — Principal Investigators Request | 1
Not completed — Withdrew Consent | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ziprasidone
Number analyzed (Participants) | 162
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.3 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72
  Male | 90

OUTCOME MEASURES:

1. Primary Outcome: Young Mania Rating Scale (YMRS) Total Score Change From Baseline
Description: YMRS: 11-item instrument with scales 0 (normal) to 4 (highest abnormal)for 7 items and 0 (normal) to 8 (highest abnormal) for 4 items. Total possible 0 - 60. Baseline is from parent study A1281132.
Time Frame: baseline and 26 Weeks; 26 Weeks Last Observation Carried Forward (LOCF)
Population: The Safety Analysis Set includes all subjects who took at least one dose of study medication in this open-label extension study. (Row: n=number subjects with observation)
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Ziprasidone
Number analyzed (Participants) | 162
score on scale
  Week 2 (n=153) | -3.8 (9.0)
  Week 6 (n=122) | -4.0 (9.1)
  Week 18 (n=76) | -6.3 (12.7)
  Week 26 (n=69) | -6.1 (11.6)
  Early Termination (n=59) | 1.5 (11.3)
  Week 26-LOCF (n=153) | -3.3 (10.7)

2. Primary Outcome: Clinical Global Impression of Severity (CGI-S) Change From Baseline
Description: CGI-S Scale:standardized assessment tool to rate severity of subject's illness; assesses investigator's impression of subject's current illness state. Change: score at observation minus score at baseline. Score: 1 (not ill at all) to 7 (among most extremely ill). Baseline = last available observation from parent double-blind study(A1281132).
Time Frame: baseline and 26 Weeks; 26 Weeks LOCF
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Ziprasidone
Number analyzed (Participants) | 162
score on scale
  Week 1 (n=159) | -0.2 (0.9)
  Week 2 (n=150) | -0.5 (1.2)
  Week 6 (n=122) | -0.4 (1.1)
  Week 10 (n=99) | -0.7 (1.3)
  Week 14 (n=85) | -0.7 (1.2)
  Week 18 (n=76) | -0.7 (1.5)
  Week 22 (n=70) | -0.8 (1.3)
  Week 26 (n=69) | -1.1 (1.4)
  Early Termination (n=48) | 0.4 (1.1)
  Week 26-LOCF (n=160) | -0.4 (1.3)

3. Primary Outcome: Incidence of Lab Abnormalities
Description: number of subjects with an abnormal lab value for those parameters with 5% or greater incidence of abnormality.
Time Frame: Week 26
Population: Total number of subjects with given laboratory test at given visit. Range: N=136-134, with the exception of Insulin (N=115)
Measure: Number; unit: participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 136
participants
  Bicarbonate (N=136) | 44
  Urine blood/Hemoglobin (N=136) | 34
  Urine ketones (N=136) | 32
  Testosterone (N=134) | 22
  Urine specific gravity (N=136) | 13
  Urine red blood cells (N=136) | 13
  Monocytes (N=134) | 9
  Triglycerides (N=136) | 10
  Urine white blood cells (N=136) | 10
  Insulin (N=115) | 8

4. Primary Outcome: Change in Low-Density Lipoprotein (LDL) Cholesterol and Fasting Cholesterol
Description: Mean Change: lab value at observation minus lab value at baseline.
Time Frame: Week 6, Week 26
Population: The Safety Analysis Set includes all subjects who took at least one dose of study medication in this open-label extension study. (Row: n= total number of subjects with at least 1 observation of the given laboratory test.)
Measure: Mean (Standard Deviation); unit: milligram /deciliter (mg/dL)
Arm/Group | Ziprasidone
Number analyzed (Participants) | 134
milligram /deciliter (mg/dL)
  LDL cholesterol Week 6 (n=113) | -7.5 (19.7)
  LDL cholesterol Week 26 (n=59) | -8.9 (19.5)
  LDL cholesterol Early Termination (n=44) | -7.6 (20.1)
  Fasting cholesterol Week 6 (n=113) | -7.7 (21.8)
  Fasting cholesterol Week 26 (n=59) | -10.3 (22.7)
  Fasting cholesterol Early Termination (n=44) | -8.6 (24.9)

5. Primary Outcome: Change in Hormones
Description: Mean Change: lab value at observation minus lab value at baseline
Time Frame: Week 6, Week 26
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: nanogram/deciliter (ng/dL)
Arm/Group | Ziprasidone
Number analyzed (Participants) | 131
nanogram/deciliter (ng/dL)
  Testosterone Week 6 (n=80) | 0.9 (84.3)
  Testosterone Week 26 (n=38) | -23.4 (112.9)
  Testosterone Early Termination (n=32) | -0.4 (61.8)
  Prolactin Week 6 (n=110) | 2.7 (13.2)
  Prolactin Week 26 (n=59) | 1.9 (8.5)
  Prolactin Early Termination (n=40) | 1.0 (11.6)
  Insulin-like growth factor Week 6 (n=95) | -19.9 (63.4)
  Insulin-like growth factor Week 26 (n=47) | -9.2 (68.1)
  Insulin-like growth factor Early Term (n=34) | -8.4 (66.5)

6. Primary Outcome: Mean Change From Baseline in Supine Systolic Blood Pressure
Description: Mean Change: vital sign value at observation minus vital sign value at baseline
Time Frame: Week 1 through Week 26
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mm Hg)
Arm/Group | Ziprasidone
Number analyzed (Participants) | 162
millimeters of mercury (mm Hg)
  Week 1 (n=155) | 0.4 (11.4)
  Week 2 (n=142) | 1.1 (10.4)
  Week 6/pre-dose (n=115) | 1.2 (9.5)
  Week 6/5-7 hours post dose (n=108) | 1.2 (9.9)
  Week 10 (n=93) | 1.4 (10.1)
  Week 14 (n=82) | -0.7 (10.1)
  Week 18 (n=74) | 0.4 (11.7)
  Week 22 (n=69) | 1.7 (10.5)
  Week 26 (n=68) | 2.9 (11.4)
  Early Termination (n=75) | 1.3 (11.8)

7. Primary Outcome: Mean Change From Baseline in Supine Diastolic Blood Pressure
Description: Mean Change: vital sign value at observation minus vital sign value at baseline
Time Frame: Week 1 through Week 26
Measure: Mean (Standard Deviation); unit: millimeters mercury (mm Hg)
Arm/Group | Ziprasidone
Number analyzed (Participants) | 162
millimeters mercury (mm Hg)
  Week 1 (n=155) | -0.5 (8.8)
  Week 2 (n=142) | 0.5 (8.7)
  Week 6/pre-dose (n=115) | 0.6 (9.7)
  Week 6/5-7 hours post dose (n=108) | 0.5 (8.8)
  Week 10 (n=93) | -0.4 (10.1)
  Week 14 (n=82) | -2.4 (8.3)
  Week 18 (n=74) | -0.6 (9.8)
  Week 22 (n=69) | -0.7 (9.4)
  Week 26 (n=68) | 1.5 (10.4)
  Early Termination (n=75) | 1.3 (8.1)

8. Primary Outcome: Mean Change From Baseline in Supine Pulse Rates
Description: Mean Change: vital sign value at observation minus vital sign value at baseline
Time Frame: Week 1 through Week 26
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Ziprasidone
Number analyzed (Participants) | 162
beats per minute
  Week 1 (n=155) | 1.4 (12.4)
  Week 2 (n=142) | 2.0 (11.7)
  Week 6/pre-dose (n=115) | -1.8 (11.6)
  Week 6/5-7 hours post dose (n=108) | 1.0 (12.3)
  Week 10 (n=93) | 1.4 (11.8)
  Week 14 (n=82) | -3.0 (12.4)
  Week 18 (n=74) | -3.5 (12.2)
  Week 22 (n=69) | -2.1 (11.7)
  Week 26 (n=68) | -3.0 (11.2)
  Early Termination (n=75) | 3.9 (13.9)

9. Primary Outcome: Mean Change From Baseline in Standing Systolic Blood Pressure
Description: Mean Change: vital sign value at observation minus vital sign value at baseline
Time Frame: Week 1 through Week 26
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Ziprasidone
Number analyzed (Participants) | 161
mm Hg
  Week 1 (n=154) | 1.4 (10.5)
  Week 2 (n=141) | 3.7 (11.7)
  Week 6/pre-dose (n=115) | 1.6 (9.6)
  Week 6/5-7 hours post dose (n=108) | 2.0 (9.5)
  Week 10 (n=93) | 2.4 (11.0)
  Week 14 (n=82) | 0.5 (11.3)
  Week 18 (n=74) | 3.1 (10.5)
  Week 22 (n=70) | 3.2 (10.0)
  Week 26 (n=68) | 3.6 (10.9)
  Early Termination (n=75) | 3.0 (11.4)

10. Primary Outcome: Mean Change From Baseline in Standing Diastolic Blood Pressure
Description: Mean Change: vital sign value at observation minus vital sign value at baseline
Time Frame: Week 1 through Week 26
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Ziprasidone
Number analyzed (Participants) | 161
mm Hg
  Week 1 (n=154) | 0.7 (9.1)
  Week 2 (n=141) | 2.0 (9.8)
  Week 6/pre-dose (n=115) | 1.4 (9.8)
  Week 6/5-7 hours post dose (n=108) | 1.2 (9.9)
  Week 10 (n=93) | 1.6 (10.8)
  Week 14 (n=82) | -0.1 (9.8)
  Week 18 (n=74) | 1.1 (8.8)
  Week 22 (n=70) | 0.5 (8.5)
  Week 26 (n=68) | 2.8 (8.3)
  Early Termination (n=75) | 3.4 (10.8)

11. Primary Outcome: Mean Change From Baseline in Standing Pulse Rates
Description: Mean Change: vital sign value at observation minus vital sign value at baseline
Time Frame: Week 1 through Week 26
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Ziprasidone
Number analyzed (Participants) | 161
beats per minute
  Week 1 (n=154) | 3.5 (14.0)
  Week 2 (n=140) | 2.9 (13.4)
  Week 6/pre-dose (n=115) | 0.3 (13.1)
  Week 6/5-7 hours post dose (n=108) | 3.8 (13.9)
  Week 10 (n=93) | 2.6 (14.5)
  Week 14 (n=82) | 0.5 (14.7)
  Week 18 (n=74) | -0.3 (12.5)
  Week 22 (n=70) | 1.2 (14.7)
  Week 26 (n=68) | -0.9 (12.9)
  Early Termination (n=75) | 4.8 (13.8)

12. Primary Outcome: Mean Change From Baseline for Body Weight
Description: Mean change; body weight value at observation minus body weight value at baseline.
Time Frame: Week 6, Week 26
Measure: Mean (Standard Deviation); unit: kilogram
Arm/Group | Ziprasidone
Number analyzed (Participants) | 162
kilogram
  Week 6 (n=119) | 1.3 (3.0)
  Week 26 (n=68) | 3.9 (5.4)
  Early Termination (n=74) | 1.4 (2.8)

13. Primary Outcome: Mean Change From Baseline for Body Mass Index (BMI) Z-Score
Description: mean change in body weight BMI -Z score calculated by subtracting median reference value of the population from observed value and dividing by standard deviation of reference population (kg/m squared). 0=no change
Time Frame: Week 6, 26, early termination
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Ziprasidone
Number analyzed (Participants) | 162
score on scale
  Week 6 (n=119) | 0.0 (0.3)
  Week 26 (n=68) | 0.1 (0.5)
  Early Termination (n=74) | 0.0 (0.3)

14. Primary Outcome: Body Mass Index (BMI) Z-score Frequency
Description: change in body weight BMI -Z score calculated by subtracting median reference value of the population from observed value and dividing by standard deviation of reference population (kg/m squared). 0=no change
Time Frame: Week 6
Measure: Number; unit: participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 162
participants
  <-4 | 0
  ≥-4 to <-3 | 0
  ≥-3 to <-2 | 0
  ≥-2 to <-1 | 0
  ≥-1 to <0 | 53
  ≥0 to <1 | 61
  ≥1 to <2 | 1
  ≥2 to <3 | 0
  ≥3 to <4 | 0
  ≥4 | 0

15. Primary Outcome: Body Mass Index (BMI) Z-score Frequency
Description: as for outcome 14
Time Frame: Week 26
Measure: Number; unit: participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 162
participants
  <-4 | 0
  ≥-4 to <-3 | 0
  ≥-3 to <-2 | 0
  ≥-2 to <-1 | 1
  ≥-1 to <0 | 27
  ≥0 to <1 | 39
  ≥1 to <2 | 1
  ≥2 to <3 | 0
  ≥3 to <4 | 0
  ≥4 | 0

16. Primary Outcome: Mean Change From Baseline for QTcF Intervals
Description: QT intervals (observed in an electrocardiogram)corrected using Fridericia's formula (QTcF). Mean change: mean change of observation minus baseline. Baseline: last available observation in the parent double-blind study.
Time Frame: Baseline to Week 26 (end of study)
Measure: Mean (Standard Deviation); unit: millisecond
Arm/Group | Ziprasidone
Number analyzed (Participants) | 162
millisecond
  Week 1 (n=152) | 4.8 (18.5)
  Week 2 (n=137) | 3.5 (17.7)
  Week 6/pre-dose (n=111) | 7.6 (17.7)
  Week 6/5-7 hours post dose (n=107) | 7.0 (18.4)
  Week 10 (n=91) | 4.3 (18.8)
  Week 14 (n=81) | 6.2 (17.4)
  Week 18 (n=73) | 7.4 (15.4)
  Week 22 (n=68) | 8.1 (16.1)
  Week 26 (n=64) | 7.1 (15.2)
  Early Termination (n=45) | 2.7 (17.0)

17. Primary Outcome: Frequency of Largest Categorical Increases in QTcF for Males
Description: QT intervals (observed in an electrocardiogram) corrected with Fridericia's Formula (QTcF). Number of subjects with corresponding categorical increase in QTcF.
Time Frame: Week 26 (end of study)
Measure: Number; unit: participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 89
participants
  ≥450 msec (millisecond ) | 0
  ≥460 msec | 0
  ≥480 msec | 0
  ≥30 msec increase | 28
  ≥60 msec increase | 0

18. Primary Outcome: Frequency of Largest Categorical Increases in QTcF for Females
Description: QT interval (observed in an electrocardiogram) corrected using Fridericia Formula (QTcF). Number of subjects with corresponding categorical increase in QTcF.
Time Frame: Week 26 (end of study)
Measure: Number; unit: participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 71
participants
  ≥450 msec (millisecond) | 3
  ≥460 msec | 0
  ≥480 msec | 0
  ≥30 msec increase | 10
  ≥60 msec increase | 2

19. Primary Outcome: Frequency of Largest Categorical Increases in QTcF - All Subjects
Description: QT intervals (observed in an electrocardiogram)corrected using Fridericia Formula (QTcF). Number of subjects with corresponding categorical increase in QTcF.
Time Frame: Week 26 (end of study)
Measure: Number; unit: participants
Arm/Group | Ziprasidone
Number analyzed (Participants) | 160
participants
  ≥450 msec (millisecond) | 3
  ≥460 msec | 0
  ≥480 msec | 0
  ≥30 msec increase | 38
  ≥60 msec increase | 2

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events are reported from time of first dose of study treatment up to 6 days after last dose of study treatment.
Description: Safety population = all randomized subjects with at least 1 dose of study treatment. An Adverse Event (AE) term may be reported as both a serious and non-serious AE, but are distinct events. AE may = serious for 1 subject and = non-serious for another subject or subject may have experienced both a serious and non-serious episode of the same event.
Arm/Group | Ziprasidone
Serious Adverse Events (participants affected / at risk) | 17/162
Other Adverse Events (participants affected / at risk) | 123/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ziprasidone (N=162)
Overdose (Injury, poisoning and procedural complications) | 1
Aggression (Psychiatric disorders) | 1
Bipolar disorder (Psychiatric disorders) | 3
Conversion disorder (Psychiatric disorders) | 1
Delusion (Psychiatric disorders) | 1
Hallucinations, mixed (Psychiatric disorders) | 1
Homicidal ideation (Psychiatric disorders) | 1
Mania (Psychiatric disorders) | 1
Negative thoughts (Psychiatric disorders) | 1
Oppositional defiant disorder (Psychiatric disorders) | 2
Self-injurious behavior (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 4
Disease progression (General disorders) | 1
Hallucination (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ziprasidone (N=162)
Abdominal pain upper (Gastrointestinal disorders) | 15
Nausea (Gastrointestinal disorders) | 13
Vomiting (Gastrointestinal disorders) | 12
Fatigue (General disorders) | 11
Dizziness (Nervous system disorders) | 12
Headache (Nervous system disorders) | 36
Sedation (Nervous system disorders) | 43
Somnolence (Nervous system disorders) | 38
Insomnia (Psychiatric disorders) | 22
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 12
Abdominal discomfort (Gastrointestinal disorders) | 11

LIMITATIONS AND CAVEATS:
The AE tables were amended to incorporate previously unreported AEs that were found during an independent audit and verified by the investigators.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.